CLINICAL TRIAL: NCT05066620
Title: An Investigator-initiated and Conducted Multicentre, Prospective, Randomised, Double-blinded Placebo-controlled Clinical Trial to Evaluate the Efficacy and Safety of Chinese Herbal Medicine in Patients With Acute Intracerebral Haemorrhage
Brief Title: Chinese Herbal Medicine in Acute INtracerebral Haemorrhage (CHAIN) Trial
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Guangzhou University of Traditional Chinese Medicine (Other)
Collaborators: The George Institute (Other)
Responsible Party: Principal Investigator, jianwen guo, MD, Professor, Guangzhou University of Traditional Chinese Medicine
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2020B1111100009
Record Dates: First submitted 2021-09-07; First posted 2021-10-04 (Actual); Last update posted 2021-10-04 (Actual); Status verified 2021-09

CONDITIONS: Intracerebral Hemorrhage
Keywords: Intracerebral haemorrhage; Functional recovery; Chinese herbal medicine; Stroke; Clinical trial
MeSH Terms: conditions — Cerebral Hemorrhage; Stroke

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): Chinese herbal medicine FYTF-919: Oral liquid 33ml TID (for patients who are unconscious or dysphagia, a dose of 25ml * Q6H will be given through nasal feeding)
  Interventions: Drug: Chinese herbal medicine FYTF-919
- Control group (Placebo Comparator): Placebo treatment: Oral liquid 33ml TID (or patients who are unconscious or dysphagia, a dose of 25ml * Q6H will be given through nasal feeding)
  Interventions: Drug: Chinese herbal medicine FYTF-919

INTERVENTIONS:
Drug: Chinese herbal medicine FYTF-919 — Oral liquid 33ml TID (for patients who are unconscious or dysphagia, a dose of 25ml * Q6H will be given through nasal feeding)
  Other Names: Chinese herbal medicine

SUMMARY:
TCM is an essential context of the ICH management in Chinese culture. Given the potential benefits of Chinese herbal medicine FYTF-919 in reducing haematoma and bleeding after acute ICH from fundamental research and small clinical studies, more reliable evidence is required to guide ICH treatment using TCM. This study aims to determine the effectiveness and safety of TCM in a larger sample of patients with moderate-severe ICH and provide evidence for TCM clinical guidelines on ICH management. The presumed mechanism of action is in promoting the reabsorption of the haematoma and perihematomal oedema in ICH.

DETAILED DESCRIPTION:
A multicentre, prospective, randomised, double-blind, placebo-controlled trial to be conducted through hospital network of investigators in China. A total of 1504 patients with ICH will be recruited from approximately 20-30 hospitals. Randomised is via a central internet-based system according to block random grouping method stratified by site, neurological severity NIHSS <15 vs ≥15), and haematoma location (basal ganglia + lobe vs thalamus + cerebellum + brain stem + ventricle) to ensure balance in key prognostic factors. Endpoint assessment will be blinded to treatment allocation. The primary aim of this study is to determine the effectiveness and safety of a Chinese herbal medicine FYTF-919 as compared to placebo on functional recovery according to Utility-weighted modified Rankin scale (UW-mRS) at 90 days after acute ICH. Secondary aims include examining whether the Chinese herbal medicine FYTF-919 leads to positive treatment effect on: 1) Utility-weighted mRS scores at 180 days; 2)Ordinal analysis of 7 levels of mRS at 28 days, 90 days and 180 days; 3) Poor prognosis, defined as mRS 4-6 points at 28 days, 90 days and 180 days; 4) NIHSS score at 7 days and 28 days; 5) Mortality rate at 28 days, 90 days and 180 days; 6) Discharge rate at 28 days; 7) EQ-5D-5L at 28days, 90 days and 180 days; 8) BI at 28 days, 90 days and 180 days; 9) The cerebral edema volume at baseline, 24 hours, 7 days, 14 days or at discharge; 10) The hematoma volume at baseline, 24 hours, 7 days, 14 days or discharge; 11) The incidence of stroke-associated pneumonia (SAP) patients; 12) Clinical pulmonary infection score (CIPS) at the onset of SAP, 3 days, and 7 days, after the occurrence of SAP; 13) Chest imaging (DR/CT), body temperature, white blood cell count, C-reactive protein (CRP), procalcitonin (PCT) blood gas analysis, and sputum culture/airway aspirate culture at the onset of SAP, 3 days, and 7 days after the occurrence of SAP; 14) Antibiotic usage among patients with SAP.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18 years;
2. Diagnosis of spontaneous ICH, confirmed by brain imaging;
3. Presentation within 48 hours of symptom onset (or last seen well);
4. Meet any of the following criteria: a) NIHSS ≥8, or b) GCS 7-14;
5. Provide written informed consent by patient (or approved surrogate);

Exclusion Criteria:

1. ICH secondary to a structural abnormality in the brain (e.g. cerebrovascular malformation, arterial aneurysm, tumour, Moyamoya disease, trauma, or previous ischaemic stroke), or secondary to presumed cerebrovascular amyloidosis, or secondary to reperfusion treatment for ischaemic stroke, or secondary to anticoagulant treatment, or secondary to antiplatelet treatment.
2. Unlikely to potentially benefit from therapy (e.g. advanced dementia) or judged by responsible treating clinician to have a high likelihood of early death irrespective of treatment;
3. Other medical illness that will interfere with outcome assessments and follow-up (e.g. known significant pre-stroke disability [modified Rankin scale {mRS} scores 4-5], advanced cancer and renal failure);
4. Known definite contraindication to the Chinese herbal medicine;
5. Women who are known to be pregnant or lactating;
6. Currently participating in another trial which would interfere with outcome assessments.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1504 (Estimated)
Dates: Start 2021-10 (Estimated); Primary Completion 2024-12 (Estimated); Study Completion 2025-01 (Estimated)

PRIMARY OUTCOMES:
Utility-weighted modified Rankin scale scores | 90 days after the treatment started
  Utility-weighted modified Rankin scale scores. The value range from 0 to 10: higher scores mean a better outcome.

SECONDARY OUTCOMES:
Utility-weighted mRS scores | 180 days after the treatment started
  Utility-weighted modified Rankin scale scores. The value range from 0 to 10: higher scores mean a better outcome.
7 levels of mRS | 28 days, 90 days and 180 days after the treatment started
  Ordinal analysis of 7 levels of mRS. The value range 0-6: higher scores mean a worse outcome.
Poor prognosis rate | 28 days, 90 days and 180 days after the treatment started
  Binary variable: 1 means mRS 4-6 points; 0 means mRS is 0-3 points.
NIHSS score | 7 days and 28 days after the treatment started
  National Institute of Health Stroke Scale Score. The value range 0-42: higher scores mean a worse outcome.
Mortality rate | 28 days, 90 days and 180 days
  Mortality rate
Discharge rate | 28 days after the treatment started
  Discharge rate
European Quality of Life 5-dimensional questionnaire (EQ-5D-5L) | 28 days, 90 days and 180 days after the treatment started
  The EQ-5D comprises five dimensions of health: mobility, ability to self-care, ability to undertake usual activities, pain and discomfort, and anxiety and depression. . EQ-5D-5L, includes five levels of severity for each dimension (no problems, slight problems, moderate problems, severe problems, and extreme problems). The value range 0-100: higher scores mean a worse outcome.
BI | 28 days, 90 days and 180 days after the treatment started
  Barthel index. The value range 0-100: higher scores mean a better outcome.
The cerebral edema volume | Baseline, 24 hours, 7 days, 14 days or at discharge
  The cerebral edema volume
The hematoma volume | Baseline, 24 hours, 7 days, 14 days or discharge
  The hematoma volume
SAP | Baseline, 24 hours, 7 days, 14 days or discharge
  The incidence of stroke-associated pneumonia patients
CPIS | The onset of SAP, 3 days and 7 days after the occurrence of SAP
  Clinical pulmonary infection score. The value range 0-12: higher scores mean a worse outcome.
Pulmonary infection | The onset of SAP, 3 days and 7 days after the occurrence of SAP
  Diagnosed by using the Chest imaging (DR/CT), body temperature, white blood cell count, C-reactive protein (CRP), procalcitonin (PCT) blood gas analysis, and sputum culture/airway aspirate culture
Antibiotic usage | The onset of SAP, 3 days and 7 days after the occurrence of SAP
  Antibiotic usage among patients with SAP

CONTACTS AND LOCATIONS:
Overall Officials: Craig Anderson, MD, Principal Investigator — The George Institute for Global Health, Australia
Locations (1):
- Guangdong Provincial Hospital of Chinese Medicine, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: Yes
Data can be shared with bona fide researchers after the publication of the main results, based on a submitted protocol to the research office of The George Institute for Global Health, Sydney Australia.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Data sharing will be available from 12 months after the publication of the main results.
Access Criteria: 1. The data sharing will be only for the purposes of health and medical research and within the constraints of the consent under which the data were originally gathered.
  2. The Custodian of the Collection will not consider any Proposals for data sharing that unblind, or potentially unblind, randomised comparisons in active / ongoing trials.
  3. Requesters should be employees of a recognised academic institution, health service organisation, commercial research organisation or from the pharmaceutical industry. Requesters must have experience in medical research.
  4. Requesters must be able to demonstrate through their peer review publications in the area of interest their ability to carry out the proposed use of the requested dataset from a Collection.
  5. The Requesters must not have a conflict of interest that may potentially influence their interpretation of any analyses.
URL: http://georgeinstitute.org.au

REFERENCES:
- [Derived] Guo J, Chen X, Wu M, Wang D, Zhao Y, Li Q, Tang G, Che F, Xia Z, Liang Z, Shi L, Jiang Q, Chen Y, Liu X, Ren X, Ouyang M, Wang B, You S, Billot L, Wang X, Liu Z, Jing H, Meng W, Tian S, Liu E, Xiang Y, Tang X, Xie T, Cui W, Zheng Y, Cao J, Zhang J, Wen Z, Huang T, Wang L, You C, Pan S, Cai Y, Lu Y, Hankey GJ, Al-Shahi Salman R, Anderson CS, Song L; CHAIN investigators. Traditional Chinese medicine FYTF-919 (Zhongfeng Xingnao oral prescription) for the treatment of acute intracerebral haemorrhage: a multicentre, randomised, placebo-controlled, double-blind, clinical trial. Lancet. 2024 Nov 30;404(10468):2187-2196. doi: 10.1016/S0140-6736(24)02261-X. Epub 2024 Nov 12. PMID 39547249